CLINICAL TRIAL: NCT00392769
Title: Phase II Study of Cetuximab (Erbitux) in Patients With Progressive or Recurrent Endometrial Cancer
Brief Title: Cetuximab in Patients With Progressive or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0211
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-08

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Progressive or Recurrent Endometrial Cancer; Cetuximab; C225; Erbitux™; IMC-C225; Epidermal growth factor receptor; EGFR; Endometrioid Tumor; Serous Tumor; Clear cell Tumor; Mixed malignant Mullerian Tumors
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab (Experimental): 400 mg/m^2 intravenous (IV) over 120 Minutes, followed by weekly infusions at 250 mg/m^2 IV over 60 minutes.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Initial Dose = 400 mg/m^2 IV Over 120 Minutes, Followed by Weekly Infusions at 250 mg/m^2 IV Over 60 Minutes.
  Other Names: C225; Erbitux™; IMC-C225

SUMMARY:
The goal of this clinical research study is to learn if cetuximab can help to control the disease in patients who have recurrent endometrial cancer.

Primary Objective:

1. To determine the overall disease control rate of cetuximab in patients with progressive or recurrent endometrial cancer.

Secondary Objectives:

1. To determine the duration of disease control, time to disease progression, and survival of this cohort of patients.
2. To determine the nature and degree of toxicity of cetuximab in this cohort of patients.
3. To correlate biologic markers with response to therapy if tissue is available.

DETAILED DESCRIPTION:
The epidermal growth factor receptor (EGFR) is a large protein that plays an important role in tumor growth. When EGFR is stimulated or "overexpressed," a series of chemical reactions happen that result in a tumor being "told" to grow. Researchers know that EGFR is overexpressed in many types of endometrial cancer. Cetuximab is designed to block this receptor, which may help to stop or slow the growth of tumors in those patients whose endometrial cancer has come back.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. If you have had some of the tests done recently, they may not need to be repeated. Your complete medical history will be recorded. You will have a physical exam, including a pelvic exam and measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate). Blood (about 2-3 teaspoons) will be drawn for routine tests, tests of your kidney and liver function, and a pregnancy test for women who are able to have children. The pregnancy test must be negative for you to be allowed to take part in this study. You will have a chest x-ray and computed tomography (CT) or magnetic resonance imaging (MRI) scans of the abdomen and pelvis (stomach and hip area) to measure the tumor.

If you are found to be eligible to take part in this study, you will receive cetuximab once a week through a needle in a vein. Each treatment cycle is 4 weeks long. In the first week of your first treatment cycle only, you will receive cetuximab over 120 minutes (2 hours). For all additional treatments, you will receive cetuximab over 60 minutes. During the infusion and for 60 minutes after the infusion ends, you will be closely watched for signs of an allergic reaction.

You will receive diphenhydramine (or a similar antihistamine) by vein, about 30-60 minutes before receiving each cetuximab infusion. This is in order to lower the risk of side effects that the study drug may cause. Your doctor may decide to lower the dose of diphenhydramine in later doses.

Before each cycle of therapy and 1 month after treatment ends, you will have a physical exam. Blood (about 2-3 teaspoons) will be drawn for routine tests. CT scans or MRI will be repeated every 2-3 cycles and at the end of treatment. If you have any tumors in your chest, a chest x-ray will be repeated every 2-3 cycles and at the end of treatment. If you have a partial or complete response (the tumor shrinks or disappears completely) or the disease is stable (where the tumor has neither grown nor shrunk), the CT or MRI will be repeated 4 weeks later to check the response.

You will be able to keep receiving additional treatment cycles as long as you are benefitting. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study.

After you have completed treatment on the study, the status of your health and the disease will be checked. Your doctor will decide how often these check-ups will occur. You may return to M. D. Anderson for these follow-up exams, or if you choose not to come in to the clinic, you will be contacted by phone to see how you are doing.

This is an investigational study. Cetuximab is commercially available and FDA approved for the treatment of colorectal cancer. Its use in the treatment of endometrial cancer in this study is experimental. Up to 40 patients will take part in this study. Up to 30 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed an approved informed consent.
2. Histologically confirmed progressive or recurrent endometrial cancer (endometrioid, serous, clear cell, mixed malignant Mullerian tumors, or mixed histology; any grade).
3. Patients must have failed at least one prior chemotherapeutic regimen for recurrent disease (does not include chemosensitizing radiation).
4. All patients must have measurable disease. Measurable disease is defined as lesions that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be > 20 mm when measured by conventional techniques, including palpation, plain x-ray, CT, and MRI, or > 10 mm when measured by spiral CT. Ascites and pleural effusions are not considered measurable disease. If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology.
5. Patients must have a Zubrod performance status of 0, 1, or 2.
6. Patients must either be not of child bearing potential or have a negative pregnancy test within 7 days of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal for greater than 12 months.
7. Patients must have a pretreatment granulocyte count (i.e., segmented neutrophils + bands) of >1,000/Fl, a hemoglobin level of >/= 9.0 gm/dL and a platelet count of >75,000/Fl.
8. Patients must have an adequate renal function as documented by serum creatinine </= 2.0 mg/dL.
9. Patients must have adequate hepatic function as documented by a serum bilirubin </= 2.5 mg/dL, regardless of whether patients have liver involvement secondary to tumor.
10. Aspartate transaminase (SGOT) must be </= 3x institutional upper limit of normal unless the liver is involved with tumor, in that case, the aspartate transaminase must be </=5 x institutional upper limit of normal.
11. Prior to beginning therapy, at least 4 weeks must have elapsed since prior chemotherapy, surgery, radiation therapy or investigational therapy. Patients receiving palliative radiation therapy are exempt from the 4 week waiting period.

Exclusion Criteria:

1. Patients who have uterine sarcomas.
2. Patients who have isolated recurrences (vaginal, pelvic, or paraaortic) that are amenable to potentially curative treatment with radiation therapy or surgery.
3. Patients with any other severe concurrent disease, which would make the patient inappropriate for entry into this study, including significant hepatic, renal, or gastrointestinal diseases.
4. Patients with a history of prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least five years.
5. Patients with active or uncontrolled systemic infection.
6. Patients with history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with an ejection fraction under 40%.
7. Patients who received prior therapy that specifically and directly targets the EGFR pathway.
8. Patients who experienced prior severe infusion reaction to a monoclonal antibody.
9. Patients who are pregnant or breast feeding.
10. Presence of clinically apparent untreated central nervous system metastases.
11. Patients with carcinomatous meningitis.
12. Patients with deep venous or arterial thrombosis (including pulmonary embolism) within 6 weeks of study entry. Patients may be on maintenance anticoagulation therapy.
13. Patients with previously documented human immunodeficiency virus (HIV) infection.
14. Patients currently receiving chemotherapy or radiation therapy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Wolf, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - New York Presbyterian Hospital-Cornell Medical Center, New York, New York
  - UT MD . Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 10, 2006 to January 25, 2010. All recruitment done in a medical clinical setting.
Period: Overall Study
Arm/Group | Cetuximab
Started | 33
Completed | 23
Not Completed | 10
Not completed — Clinical Deterioration | 9
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab
Number analyzed (Participants) | 33
Age Continuous [Median (Full Range); unit: years] | 63 [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Disease Control Rate
Description: Overall disease control rate also called the Clinical Benefit Response (CBR) is defined as Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) evaluated within 8 weeks (CR or PR) and 12 weeks (SD) of initial treatment, using Bayesian design.
Time Frame: Overall disease control rate (CR + PR + SD) evaluated within 8 weeks (CR or PR) and 12 weeks (SD) of initial treatment.
Population: There were ten inevaluable participants (completing less than 1 cycle).
Measure: Number; unit: percentage of participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 23
percentage of participants | 17

ADVERSE EVENTS:
Time Frame: 3 years and 5 months
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 23/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=33)
Rash (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 13
Nausea (Gastrointestinal disorders) | 1
Headache (General disorders) | 3
Pain (all sites) (General disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=33)
Rash (Skin and subcutaneous tissue disorders) | 24
Fatigue (General disorders) | 21
Constipation (Gastrointestinal disorders) | 8
Headache (General disorders) | 8
Nausea (Gastrointestinal disorders) | 11
Pain (all sites) (General disorders) | 8
Vomiting (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No